CLINICAL TRIAL: NCT03708978
Title: Development of Artificial Intelligence System for Detection and Diagnosis of Breast Lesion Using Mammography
Status: Completed | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Peking University (Other)
Responsible Party: Principal Investigator, Sun Ying-Shi, Chairman of Dept.Radiology, Peking University Cancer Hospital & Institute
Other Study IDs: BCA-AI
Record Dates: First submitted 2018-04-17; First posted 2018-10-17 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Women With Breast Cancer
MeSH Terms: interventions — Mammography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — If a subject is diagnosed with BI-RAD4/5, she will receive pathological biopsy. The tissue sample from biopsy will be used to give a definitive malignant or benign diagnosis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mammography group: women who receives mammography because of suspected breast lesion(s)
  Interventions: Diagnostic Test: mammography

INTERVENTIONS:
Diagnostic Test: mammography — When a woman comes to the clinic to receive mammography. Then a radiologist will give a BI-RADS classification after reviewing the images. If a BI-RADS 4/5 is obtained, the woman will receive pathological biopsy to ensure there is a benign or malignant lesion. If a BI-RADS 3 is obtained, the woman will be followed up by a half-year interval until two year after the first mammography. At each follow up, she will receive mammography. If a BI-RADS 4/5 is obtained at follow up, she will receive pathological biopsy; if a BI-RADS 1/2/3 is obtained at follow up, she will be followed up by a half-year interval until two year. If a BI-RADS 1/2 is obtained at the first mammography, the woman will receive a second mammography after two year. During the study period, breast examination and results will be recorded for every subject. Radiologists will give the diagnosis with and without AI support.

SUMMARY:
This project aims to establish a comprehensive artificial intelligence system for detecting and qualitative diagnosing breast lesions. Mammary images will be used to construct a diagnosis method based on deep learning. The system is proposed to automatically analyze the type of mammary glands, automatically identify and mark all breast lesions on the mammography images, provide the malignancy probability judgment of the lesions, the BI-RADS classification and the clinical suggestion, and also automatically generate the structured diagnosis report.

DETAILED DESCRIPTION:
This is a multi-center study.The project contains a retrospective part(3000 samples anticipated) and a prospective part(7000 samples anticipated). In the retrospective part, investigators collected subjects with mammary images to design the deep learning method and construct a detective and diagnostic model for breast lesions. In the prospective part, investigators validate the accuracy of the constructed deep learning method, and established artificial intelligence system focusing on mammary diagnosis. Investigators will also explore the application pattern of the artificial intelligence system in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* the X-ray images of the breast were complete
* the results of pathological diagnosis or more than 2 years of mammography follow-up were available
* subject signs informed consent(this item was only for prospective study cases)

Exclusion Criteria:

* there exists pathological diagnosis of breast lesions when receiving mammography
* there lacks pathological diagnosis or 2 years of mammography follow-up
* subject withdraws(this item was only for prospective study cases)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with suspected Breast Lesion
Sampling Method: Probability Sample
Enrollment: 5809 (Actual)
Dates: Start 2018-04-05 (Actual); Primary Completion 2020-05-04 (Actual); Study Completion 2020-05-04 (Actual)

PRIMARY OUTCOMES:
benign-malignant diagnosis accuracy | from the first mammography to pathological result obtained(an average of 3 weeks if mammography BI-RADS 4 or 5 obtained)
  the accuracy of the AI model, radiogist with AI support, radiologist alone for binary diagnosis of a benign or malignant breast lesion according to pathology. If either one mammography of BI-RADS 4/5 in the first examination or during the two year' follow up examination is obtained,a pathological examination is performed, the lesion is judged benign or malignant according to pathological results.
benign-malignant diagnosis accuracy | from the first mammography to 2-year-after mammography
  the accuracy of the AI model, radiogist with AI support, radiologist alone for binary diagnosis of a benign or malignant breast lesion according to follow up. If a 2-year mammography of BI-RADS 1/2/3 is obtained, the lesion is considered benign. If either one mammography of BI-RADS 4/5 during the two year is obtained,a pathological examination is performed to ensure the benign or malignant lesion

SECONDARY OUTCOMES:
lesion detection accuracy | from the first mammography to radiologist diagnosis (within 3 days after the mammography taken)
  the detection rate of the constructed deep learning method for detecting benign or malignant breast lesion according to radiologist's subjective diagnosis or follow up as reference. If a radiologist suggests existence of a lesion at the first mammography or at each follow-up mammography during the 2-year period, it is considered that a lesion exists

CONTACTS AND LOCATIONS:
Overall Officials: Ying-Shi Sun, Professor, Study Chair — Peking University Cancer Hospital & Institute
Locations (8):
- China (8):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chao Yang Women and Children's Health Hospital, Beijing, Beijing Municipality
  - Beijing Da Xing People's Hospital, Beijing, Beijing Municipality
  - Beijing Hang Tian Centre Hospital, Beijing, Beijing Municipality
  - Beijing Nan Jiao Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Shi Jing Shan Hospital, Beijing, Beijing Municipality
  - Beijing Shun Yi Qu Hospital, Beijing, Beijing Municipality
  - Beijing Shun Yi Woman and Children Health Hospital, Beijing, Beijing Municipality

IPD SHARING:
Plan to Share IPD: No